CLINICAL TRIAL: NCT02729675
Title: Innovative Approaches to Increase F&V Intake Thru Worksites: The Fresh Initiative
Brief Title: Innovative Approaches to Increase F&V Intake Thru Worksites
Acronym: Good to Go
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Kim Gans, Principal Investigator/Adjunct Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01CA133396 (NIH)
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Food Habits; Eating Behavior
Keywords: fruit & vegetable, market, education, worksite, food access
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Access Intervention (Experimental): Worksites in this condition received weekly Fruit and Vegetable markets
  Interventions: Other: Access Intervention
- Enhanced Intervention (Experimental): Worksites in this condition received weekly Fruit and Vegetable markets and Educational Interventions including Campaigns, Newsletters, DVDs, A Website, and Chef Demonstrations
  Interventions: Other: Access Intervention; Behavioral: Enhanced Intervention
- Comparison Intervention (Active Comparator): Worksites in this condition received Stress and Physical Activity Interventions
  Interventions: Behavioral: Comparison Behavioral Intervention

INTERVENTIONS:
Other: Access Intervention — The 7 worksites in this arm received year-round, weekly mobile F&V markets (Fresh To You - FTY) selling local and non-local fresh produce at or below local supermarket prices. The markets carried 50 to 70 different produce items and were held both indoors and outdoors depending on the weather and worksite preference. When held indoors, F&V were sold in a cafeteria or other highly trafficked area. In good weather, the markets were held outside on the worksite property in a retrofitted a car trailer. Each market lasted two hours. On average, FTY prices were 15% to 25% lower than local retail supermarket prices. Signs, posters, email blasts and flyers advertised the markets. The FTY intervention at each worksite began with a Kick-Off event, which included the first FTY market. Each employee who attended the first market received a large, reusable shopping bag with the FTY logo on it and a freezer pack to keep F&V fresh.
  Other Names: Fresh to You Fruit and Vegetable Mobile Market Intervention
  Arms: Access Intervention; Enhanced Intervention
Behavioral: Enhanced Intervention — The 7 worksites in this arm received the Access intervention described above as well as set of educational/behavioral interventions. At the Kick-Off, employees received the first month's newsletter and an educational digital video disk (DVD) in the reusable shopping bag. They also received a chef-run cooking demonstration/taste-testing along with recipes and information about the upcoming intervention activities. Intervention activities included two 6-week campaigns (Just Add Two and Choose Color, Choose Health); a 90 minute DVD with cooking demonstrations about preparing quick, healthy inexpensive meals and unusual F&V; a two-page, full-color newsletter distributed monthly; Food demonstrations/tastings delivered once a month by chefs including an easy to prepare, F&V-based recipe; a total of 12 recipe handouts that correlated with the monthly cooking demonstration; a Good to Go website; and a project bulletin board.
  Other Names: Educational plus Access Intervention
  Arms: Enhanced Intervention
Behavioral: Comparison Behavioral Intervention — Brown University contracted with the Greater Providence Young Men's Christian Association (YMCA) to provide a physical activity and stress reduction intervention at the 7 worksites in the comparison group. Two, six-week campaigns were developed jointly by the Brown study team and YMCA staff. These campaigns followed the same format as the enhanced intervention group campaigns and were provided during the same time periods as those at the enhanced intervention sites. Everyone who participated in the campaigns also received a free, 6-week membership to the YMCA.
  Other Names: Attention Placebo Control
  Arms: Comparison Intervention

SUMMARY:
The purpose of this project is to study the efficacy of a delivery system to offer fresh fruits and vegetables (F&V) at discount prices for purchase at worksites in conjunction with educational interventions on increasing employees' F&V consumption in comparison to an intervention receiving fruit and vegetable markets alone or a comparison intervention.

DETAILED DESCRIPTION:
"Good to Go" (GTG) is a cluster randomized trial, which is studying the efficacy of innovative multi-level worksite interventions including educational/behavioral interventions and/or a fruit and vegetable (F&V) market at the worksite to improve F&V intake of employees. The hypothesis is that providing convenient, inexpensive access to F&V at the workplace through a F&V market will increase the availability of F&V at the workplace as well as at home and increase F&V intake of the employee. However, because it is unclear if improving F&V access and availability alone is adequate to increase F&V intake, the investigators will test the efficacy of the F&V delivery intervention alone and in combination with a promotional/educational intervention delivered at the worksite. The efficacy of these innovative interventions will be tested during a cluster randomized trial with 21 worksites to determine which interventions are most efficacious in increasing F&V consumption.

The primary specific aims of this proposed research are to employ a cluster randomized trial to study the efficacy of delivering fresh F&V at reduced prices for purchase at worksites (access intervention); the F&V delivery intervention paired with educational interventions to change informational and social environments at the worksite (enhanced intervention); and a comparison intervention acting as an attention placebo. The study will compare the efficacy of the Access intervention and the enhanced intervention with the comparison Arm and will also compare the efficacy of the Access intervention to the Enhanced intervention.

ELIGIBILITY:
Inclusion Criteria:

* works at least 25 hours per week at the worksite
* is on-site at least half of every day shift during the week
* reads and understands English.

Exclusion Criteria:

* has a medical condition that would prevent consumption of most fruits and vegetables,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1804 (Actual)
Dates: Start 2010-09; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Intake | Baseline, 6 and 12 months
  Measured by National Cancer Institute Eating at America's Table All Day Screener
Change in Fruit and Vegetable Intake | Baseline, 6 and 12 months
  Two-Item Cup F&V intake screener

SECONDARY OUTCOMES:
Change in fruit and vegetable eating behaviors | Baseline, 6 and 12 months
  F&V habits questions

CONTACTS AND LOCATIONS:
Overall Officials: KIM Gans, Principal Investigator — Brown University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Risica PM, Gorham G, Dionne L, Nardi W, Ng D, Middler R, Mello J, Akpolat R, Gettens K, Gans KM. A multi-level intervention in worksites to increase fruit and vegetable access and intake: Rationale, design and methods of the 'Good to Go' cluster randomized trial. Contemp Clin Trials. 2018 Feb;65:87-98. doi: 10.1016/j.cct.2017.12.002. Epub 2017 Dec 12. PMID 29242108